CLINICAL TRIAL: NCT05605899
Title: An Adaptive Phase 3, Randomized, Open-Label, Multicenter Study to Compare the Efficacy and Safety of Axicabtagene Ciloleucel Versus Standard of Care Therapy as First-Line Therapy in Subjects With High-Risk Large B-Cell Lymphoma (ZUMA-23)
Brief Title: Study to Compare Axicabtagene Ciloleucel With Standard of Care Therapy as First-line Treatment in Participants With High-risk Large B-cell Lymphoma
Acronym: ZUMA-23
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Organization: Gilead Sciences (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KT-US-484-0136; 2022-501489-24-00 (Other: European Medicines Agency)
Record Dates: First submitted 2022-10-31; First posted 2022-11-04 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: High-risk Large B-cell Lymphoma (LBCL)
MeSH Terms: interventions — axicabtagene ciloleucel; Cyclophosphamide; fludarabine; Etoposide; Rituximab; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Axicabtagene Ciloleucel (Experimental): Participants will receive cyclophosphamide 500 mg/m^2/day intravenously (IV) and fludarabine 30 mg/m^2/day IV lymphodepletion chemotherapy for 3 days followed by axicabtagene ciloleucel administered as a single IV infusion at a target dose of 2 x 10^6 anti-cluster of differentiation (CD)19 chimeric antigen receptor (CAR) transduced autologous T cells/kg on Day 0.
  Interventions: Biological: Axicabtagene Ciloleucel; Drug: Cyclophosphamide; Drug: Fludarabine
- Standard of Care Therapy (Active Comparator): Participants will receive the investigator's choice of one of the following therapies/dosing schedules:
  * Rituximab plus cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP) for a total of 6 cycles (21-day cycle)
    * Rituximab 375 mg/m^2 on Day 1
    * Cyclophosphamide 750 mg/m^2 on Day 1
    * Doxorubicin 50 mg/m^2 on Day 1
    * Vincristine 1.4 mg/m^2 (maximum 2 mg) on Day 1
    * Prednisone 40 mg/m^2 on Day 1 through Day 5
  * Dose-adjusted etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, and rituximab (DA-EPOCH-R) for a total of 6 cycles (21-day cycle)
    * Rituximab 375 mg/m^2 on Day 1
    * Etoposide 50 mg/m^2 on Days 1 to 4
    * Doxorubicin 10 mg/m^2 on Days 1 to 4
    * Vincristine 0.4 mg/m^2 on Days 1 to 4
    * Cyclophosphamide 750 mg/m^2 on Day 5
    * Prednisone 60 mg/m^2 twice daily on Days 1 to 5
  Interventions: Drug: Cyclophosphamide; Drug: Etoposide; Drug: Rituximab; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone

INTERVENTIONS:
Biological: Axicabtagene Ciloleucel — A single infusion of chimeric antigen receptor (CAR)-transduced autologous T cells
  Other Names: Yescarta®; Axi-cel
  Arms: Axicabtagene Ciloleucel
Drug: Cyclophosphamide — Administered intravenously
Drug: Fludarabine — Administered intravenously
  Arms: Axicabtagene Ciloleucel
Drug: Etoposide — Administered intravenously
  Arms: Standard of Care Therapy
Drug: Rituximab — Administered intravenously
  Arms: Standard of Care Therapy
Drug: Doxorubicin — Administered intravenously
  Arms: Standard of Care Therapy
Drug: Vincristine — Administered intravenously
  Arms: Standard of Care Therapy
Drug: Prednisone — Administered orally
  Arms: Standard of Care Therapy

SUMMARY:
The goal of this clinical study is to compare the study drug, axicabtagene ciloleucel, versus standard of care (SOC) in first-line therapy in participants with high-risk large B-cell lymphoma.

DETAILED DESCRIPTION:
Five years after randomization, participants who have received axicabtagene ciloleucel will transition to a separate long-term follow-up study (study KT-US-982-5968) to complete the remainder of the 15-year follow-up assessments.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed large B cell lymphoma (LBCL) based on 2016 World Health Organization (WHO) classification by local pathology lab assessment, including of the following:

  * Diffuse large B-cell lymphoma (DLBCL), not otherwise specified (NOS)
  * High-grade B-cell lymphoma (HGBL)
* Note: Transformed DLBCL from follicular lymphoma or from marginal zone lymphoma is eligible if no prior treatment with anthracycline-containing regimen.
* High-risk disease defined as an International Prognostic Index (IPI) score of 4 or 5 at initial diagnosis.
* Have received only 1 cycle of rituximab plus chemotherapy (R-chemotherapy).
* Adequate bone marrow, renal, hepatic, pulmonary, and cardiac function.
* Females of childbearing potential must have a negative serum or urine pregnancy test.

Key Exclusion Criteria:

* The following WHO 2016 subcategories by local assessment:

  * T-cell/histiocyte-rich LBCL
  * Primary DLBCL of the central nervous system (CNS)
  * Primary mediastinal (thymic) LBCL
  * B-cell lymphoma, unclassifiable, with features intermediate between DLBCL and classical Hodgkin lymphoma
  * Burkitt lymphoma
  * History of Richter's transformation of chronic lymphocytic leukemia
* Presence of detectable cerebrospinal fluid (CSF)-malignant cells, brain metastases, or a history of CNS involvement of lymphoma.
* Presence of cardiac lymphoma involvement.
* Any prior treatment for LBCL other than the 1 cycle of R-chemotherapy.
* History of severe immediate hypersensitivity reaction to any of the agents used in this study.
* Presence of CNS disorder. History of stroke, transient ischemic attack, or posterior reversible encephalopathy syndrome (PRES) within 12 months prior to enrollment.
* History of acute or chronic active hepatitis B or C infection.
* Positive for human immunodeficiency virus (HIV) unless taking appropriate anti-HIV medications, with an undetectable viral load by PCR and with a cluster of differentiation 4 (CD4) count > 200 cells/uL.
* Medical conditions or residual toxicities from prior therapies likely to interfere with assessment of safety or efficacy of study treatment. Please refer to protocol for further details.
* History of clinically significant cardiac disease within 12 months before enrollment.
* History of any medical condition requiring maintenance systemic immunosuppression/systemic disease modifying agents within the last 2 years.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-02-10 (Actual); Primary Completion 2031-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Event-free Survival (EFS) by Blinded Central Assessment | Up to 5 years
  EFS, is defined as the time from randomization to the earliest occurrence of death due to any cause, disease progression/relapse, initiation of any non-protocol specified subsequent new lymphoma therapy for the treatment of residual disease or Biopsy-proven residual disease at the Month 6 disease assessment or later, regardless of whether subsequent new lymphoma therapy is initiated or not.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) by Blinded Central Assessment | Up to 5 years
  PFS is defined as the time from randomization to disease progression or death due to any cause.
Overall Survival | Up to 5 years
  OS is defined as the time from randomization to death due to any cause.
PFS by Investigator Assessment | Up to 5 years
  PFS is defined as the time from randomization to disease progression or death due to any cause.
Complete Response (CR) Rate by Blinded Central Assessment | Up to 5 years
  CR rate is defined as the proportion of participants who have achieved CR per Lugano classification after treatment completion and prior to subsequent new off protocol anti-lymphoma therapy.
Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Deaths | First dose date up to 5 years plus 30 days
Percentage of Participants Experiencing Clinically Significant Changes in Safety Laboratory Values | First dose date up to 5 years plus 30 days
Change From Baseline in the European Organisation for Research and Treatment of Cancer-Quality of Life Questionnaire-30 (EORTC QLQ-C30) Score | Baseline, Month 18
  The EORTC-QLQ-C30 is a multi-item questionnaire measuring the following content: five (5) multi-item functional scales, three (3) multi-item symptom scales, six (6) symptom single-item scales, one (1) global health status scale, and one (1) global health-related quality of life (HRQoL). Each scale is measured from 0 to 100 after a linear transformation. Higher scores for functioning scales and for the Global Health Status or Global HRQoL scales indicate a higher level of functioning and a better HRQoL respectively, whereas higher scores in symptom scales represent a higher level of symptoms.
Change From Baseline in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Non-Hodgkin Lymphoma High Grade Module (EORTC QLQ-NHL-HG29) Score | Baseline, Month 18
  The EORTC QLQ-NHL-HG29 is a 29-item patient-reported assessment measuring patients' high-grade NHL-specific symptoms and functioning. The 29 items assess symptom burden due to disease and/or treatment, fatigue/physical condition, neuropathy, emotional impacts, and worries/fears health and functioning. Each scale is measured from 0 to 100 after a linear transformation. Higher scores for functional scales indicate a higher level of functioning and a better HRQoL, whereas higher scores in symptom scales represent a higher level of symptoms.
Change From Baseline in the European Quality of Life Five Dimensions Five Levels Questionnaire (EQ-5D-5L) Score | Baseline, Month 18
  The EQ-5D-5L questionnaire is a generic measure of health status that provides a simple descriptive profile and a single index value. The EQ-5D-5L comprises 2 components: a questionnaire covering 5 dimensions and a tariff of values based upon direct valuations of health states using a visual analog scale (VAS). Rating gets recorded on a vertical VAS in which the endpoints are labeled best imaginable health state is 100 (on the top) and worst imaginable health state is 0 (on the bottom). Higher scores of EQ VAS indicate better health.

CONTACTS AND LOCATIONS:
Overall Officials: Kite Study Director, Study Director — Kite, A Gilead Company
Locations (90):
- United States (37):
  - University of Alabama Hospital, Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic, Phoenix, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of California Los Angeles (UCLA), Los Angeles, California
  - Stanford Cancer Institute, Palo Alto, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - The University of Kansas Hospital, Westwood, Kansas
  - Norton Cancer Institute, St. Matthews Campus, Shelbyville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of MD Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Cancer Center Outpatient Pharmacy, Rochester, Minnesota
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Weill Cornell Medical College - NewYork Presbyterian Hospital, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Novant Health Cancer Institute- Hematology, Charlotte, North Carolina
  - Oncology Hematology Care Clinical Trials, LLC, Cincinnati, Ohio
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Prisma Health Cancer Institute, Greenville, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Henry-Joyce Cancer Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The University of Texas, MD Anderson Cancer Center, Houston, Texas
  - Intermountain LDS Hospital/Blood and Marrow Transplant/ Acute Leukemia Program, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Australia (3):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Royal Brisbane and Women's Hospital, South Brisbane, Queensland
  - Peter MacCallum Cancer Center, Melbourne, Victoria
- Austria (4):
  - Medizinische Universität Innsbruck, Innsbruck
  - Zuniklinikum Salzburg, Landeskrankenhaus, Universitatsklinik fur Innere Medizin III der PMU, Salzburg
  - Universitätsklinikum St. Pölten, Sankt Pölten
  - Medizinische Universität Wien (AKH Wien, Medical University Vienna and General Hospital Vienna), Vienna
- Canada (3):
  - Jewish General Hospital, Montreal
  - The Ottowa Hospital- General Campus, Ottawa
  - Princess Margaret Cancer Centre, Toronto
- France (9):
  - CHU Bordeaux-Hopital Haut-Leveque, Bordeaux
  - Centre Leon Berard, Cedex Lyon 08
  - CHU Dijon, Dijon
  - Hopital Claude Huriez CHU Lille, Service Maladies du sang, Lille
  - Hopital Saint Eloi, Montpellier
  - Centre Hospitalier Universitaire de Nice, Nice
  - Hopital Henri MONDOR, APHP, Paris
  - CHU Pontchaillou, Rennes
  - Centre Hospitalier Universitaire(CHU) de Toulouse, Toulouse
- Germany (5):
  - Helios Klinikum Berlin-Buch, Berlin
  - Charite Universitaetsmedizin Berlin, Berlin
  - Universitätsklinikum bonn, medizinische klinik III, Bonn
  - Uniklinikum Duesseldorf, Klinik fuer Haematologie, Onkologie und klinische Immunologie, Düsseldorf
  - Universitätsklinik Erlangen, Erlangen
- Italy (7):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna
  - ASST Degli Spedali Civili di Brescia, Brescia
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliera di Perugia - Ospedale S. Maria della Misericordia, Perugia
  - Grande Ospedale Metropolitano Bianchi Melacrino Morelli, Reggio Calabria
  - Universita Cattolica del Sacro Cuore, Rome
  - IRCCS Istituto Clinico Humanitas, Rozzano
- Japan (5):
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto
  - Tohoku University Hospital, Miyagi
  - Osaka University Hospital, Osaka
  - Juntendo University Hospital, Tokyo
  - Tokyo Metropolitan Komagome Hospital, Tokyo
- Netherlands (5):
  - Academisch Medisch Centrum, Amsterdam
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Maastricht Universitair Medisch Centrum, Maastricht
  - Universitair Medisch Centrum Utrecht, Utrecht
- Portugal (3):
  - Centro Hospitalar Universitario Lisboa Norte, E.P.E. - Hospital de Santa Maria, Lisbon
  - Instituto Portugues de Oncologia de Lisboa Francisco Gentil - E.P.E., Lisbon
  - Instituto Portugues de Oncologia do Porto Francisco Gentil, E.P.E., Porto
- Spain (7):
  - Institut Catala d'Oncologia, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
- United Kingdom (2):
  - Addenbrookes Hospital (Cambridge University Hospitals NHS Foundation Trust), Birmingham
  - University Hospitals Southampton, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — http://www.gileadclinicaltrials.com/study/?id=KT-US-484-0136